CLINICAL TRIAL: NCT05584059
Title: Pai.ACT: A Deep-Learning Mental Health Advisory System Using Acceptance and Commitment Therapy for Parents of Children With Special Healthcare Needs (Phase I)
Brief Title: Pai.ACT Programme for Parents of Children With Special Healthcare Needs - Phase I
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Hong Kong Association of Youth Department (Unknown); Hong Kong Christian Service (Other); Hong Kong Federation of Youth Groups (Unknown); Hong Kong School Nurse Association (Unknown); Hong Kong Young Women's Christian Association (Other); Yang Memorial Methodist Social Service (Other)
Responsible Party: Principal Investigator, Yuen Yu CHONG, Assistant Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ITB/FBL/6033/21/P
Record Dates: First submitted 2022-10-14; First posted 2022-10-18 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Neurodevelopmental Disorders; Attention Deficit Hyperactivity Disorder; Autism Spectrum Disorder; Development Delay; Chronic Disease
Keywords: Focused Acceptance and Commitment Therapy; Special health care needs; Mobile App; Machine Learning
MeSH Terms: conditions — Neurodevelopmental Disorders; Attention Deficit Disorder with Hyperactivity; Autism Spectrum Disorder; Learning Disabilities; Chronic Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FACT Group (Experimental): 4-6 weeks of 45-60 minute individual-based Focused Acceptance and Commitment Therapy (FACT) counselling sessions delivered via video-conferencing format or face-to-face
  Interventions: Behavioral: Focused Acceptance and Commitment Therapy

INTERVENTIONS:
Behavioral: Focused Acceptance and Commitment Therapy — This is an individual-based FACT counselling programme which composes of 4-6 sessions on a weekly basis (45-60mins/session). All the sessions are delivered by a trained FACT interventionist via either video-conferencing (e.g., Zoom or Windows Teams) or face-to-face format. The programme aims to increase the psychological flexibility of the parent, so that he/she is able to (i) experience the present moment and take perspective on self (i.e., Awareness); (ii) detach the distressing private experiences and associated rules and to take a non-judgemental, accepting stance toward the painful experiences (i.e., Openness) and (iii) exhibits strong connection with values and commit to values-consistent actions. The trained interventionist will use different ACT strategies in these sessions, including ACT metaphors, experiential exercises, guided mindfulness exercises, guided imagery exercises and values clarification exercises to reinforce the above principles.

SUMMARY:
This study aims to determine the feasibility, acceptability and potential efficacy of an individual, video-conferencing based Focused Acceptance and Commitment Therapy (FACT) on the mental well-being of parents of children with Special Health Care Needs(SHCN). The study also aims to explore the experience of parents after participating in the individual-based FACT sessions offered by the trained FACT interventionists.

DETAILED DESCRIPTION:
Parents of children with Special Health Care Needs (SHCN) have always been under tremendous pressure to care for their children. They have been experiencing significant caregiving difficulties, such as scheduling and accompanying multiple follow-ups for rehabilitation and functional recovery and managing the child's symptoms and problematic behaviours. With the strike of COVID-19, these parents' stress may even be exacerbated due to the lockdown measures. Children's needs become more demanding with the suspension of the usual care services. Parenting stress has been known to affect parent-child interactions and increase negative parenting behaviours such as harsh, permissive or neglecting parenting impairing the parent's capacity to respond to the demands of the child's illness, which may, in turn, exacerbate the child's health problem and well-being. Recent evidence has advocated the efficacy of Acceptance and Commitment Therapy (ACT) on mental health in different population groups, including healthy individuals, parents, children and those with mental health problems. To increase the reach of ACT and overcome the plausible disruptions of mental health services arising from the pandemic, the study proposes to use an innovative intervention approach, that is a brief version of ACT (Focused ACT), delivered by trained FACT interventionists in individual-based, video-conferencing format. The conversation data between the parent and the interventionist will be further analyzed for developing a Deep-Learning Mental Health Advisory System in the second phase of the Pai.ACT project. This study aims to determine the feasibility, acceptability and potential efficacy of an individual, video-conferencing-based Focused Acceptance and Commitment Therapy (FACT) on the mental well-being of parents of children with Special Health Care Needs(SHCN). The study also aims to explore the experience of parents after participating in the individual-based FACT sessions offered by the trained FACT interventionists.

ELIGIBILITY:
Inclusion Criteria:

* Cantonese-speaking Hong Kong residents
* living together with the child who is at preschool/school-age (3-9 years old)
* adopt the responsibility of taking care of the child,
* has daily access to their iPhone and Android smartphones.

In addition, potential eligible parents who respond "yes" to any of the five validated screening questions in the Children with Special Health Care Needs (SHCN) Screener (see https://www.childhealthdata.org/docs/cshcn/technical-summary-of-cshcn-screener.pdf) will then be asked the associated follow-up questions to determine whether the child possesses physical, neurodevelopmental/emotional problem(s) that has lasted for at least 12 months. Only children with a positive response(s) to ≥ 1 item in each of the associated follow-up questions will be classified as children with SHCN.

Exclusion Criteria:

* Parents with severe mental illness or developmental disabilities which impaired their ability to comprehend the content of the programme will be excluded.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Parental depressive symptoms | Change from baseline assessment to immediate post-assessment
  The Patient Health Questionnaire (PHQ-9, 9-item, 4-point Likert scale) will be used to assess the frequency of the parents experiencing depressive symptoms in the past two weeks. The Chinese version of the PHQ-9 has demonstrated good internal consistency reliability (Cronbach's alpha = 0.86) and a 2-week test-retest correlation coefficient.
Parental anxiety symptoms | Change from baseline assessment to immediate post-assessment
  The Generalized Anxiety Disorder-7 (GAD-7, 7-item, 4-point Likert scale) will be used to measure the severity of anxiety symptoms. The Chinese version of the GAD-7 demonstrated good reliability and validity with a Cronbach's coefficient of 0.91.
Parental Stress | Change from baseline assessment to immediate post-assessment
  The Parental Stress Scale (PSS, 16-item, 5-point scale) will be used to assess parenting stress. A higher score represents a higher level of parental stress. The Chinese version of the PSS has demonstrated acceptable psychometric properties and is therefore suitable for use by researchers to assess the parental stress levels of Chinese parents.

SECONDARY OUTCOMES:
Parental Psychological Flexibility | Change from baseline assessment to immediate post-assessment
  The PsyFlex (6-item 5-point Likert Scale) will assess all the six therapeutic processes of Acceptance and Commitment Therapy (ACT). Each item refers to one of the core skills that ACT focuses on when developing psychological flexibility and well-being. The score is then interpreted such that higher scores represent higher psychological flexibility.

CONTACTS AND LOCATIONS:
Overall Officials: Yuen Yu Chong, PhD, Principal Investigator — Chinese University of Hong Kong
Locations (5):
- Hong Kong (5):
  - Hong Kong Christian Service, Hong Kong
  - Hong Kong Federation of Youth Groups, Hong Kong
  - Hong Kong School Nurse Association, Hong Kong
  - Hong Kong Young Women's Christian Association, Hong Kong
  - Yang Memorial Methodist Social Service, Hong Kong